CLINICAL TRIAL: NCT02942771
Title: A Phase 1b, Double-Blind, Randomized, Placebo-Controlled Multiple Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetic Profile of TT301/MW189 Administered Intravenously to Healthy Volunteers
Brief Title: A MAD Study of TT301/MW189 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Linda Van Eldik (Other)
Collaborators: Duke Clinical Research Institute (Other); Alzheimer's Association (Other)
Responsible Party: Sponsor-Investigator, Linda Van Eldik, Sponsor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TT301/MW189 Phase 1b
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Results first posted 2020-06-02 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Healthy Adult Volunteers
MeSH Terms: interventions — TT-301

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 - TT301/MW189 (Experimental): TT301/MW189 0.075 mg/kg IV (or matched placebo). Each subject will receive 1 dose level of study drug twice daily (bid) on Days 1 through 5, inclusive
  Interventions: Drug: 0.075mg/kg TT301/MW189
- Cohort 2 -TT301/MW189 (Experimental): TT301/MW189 0.15 mg/kg IV (or matched placebo). Each subject will receive 1 dose level of study drug twice daily (bid) on Days 1 through 5, inclusive
  Interventions: Drug: 0.15mg/kg TT301MW189
- Cohort 3- TT301/MW189 (Experimental): TT301/MW189 0.25 mg/kg IV (or matched placebo). Each subject will receive 1 dose level of study drug twice daily (bid) on Days 1 through 5, inclusive
  Interventions: Drug: 0.25mg/kg TT301/MW189
- Cohort 4- TT301/MW189 (Experimental): TT301/MW189 0.30 mg/kg IV (or matched placebo). Each subject will receive 1 dose level of study drug twice daily (bid) on Days 1 through 5, inclusive
  Interventions: Drug: 0.30mg/kg TT301/MW189
- Placebo (Placebo Comparator): No drug intervention.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 0.075mg/kg TT301/MW189 — 0.075 mg/kg IV twice daily on Days 1 through 5
  Other Names: TT301/MW189
  Arms: Cohort 1 - TT301/MW189
Drug: 0.15mg/kg TT301MW189 — 0.15 mg/kg IV twice daily on Days 1 through 5
  Other Names: TT301/MW189
  Arms: Cohort 2 -TT301/MW189
Drug: 0.25mg/kg TT301/MW189 — 0.25 mg/kg IV twice daily on Days 1 through 5
  Other Names: TT301/MW189
  Arms: Cohort 3- TT301/MW189
Drug: 0.30mg/kg TT301/MW189 — 0.30 mg/kg IV twice daily on Days 1 through 5
  Other Names: TT301/MW189
  Arms: Cohort 4- TT301/MW189
Drug: Placebo — 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
The purpose of this Study is to find out whether an investigational drug is safe and well tolerated. MW189 is being studied as a possible short-term treatment for people with different types of brain injury. MW189 has previously been given to healthy human volunteers as a single dose, and there were no significant problems or bad effects in people who received the Study drug. However, before it can be tested in people with brain injury, it is important to test MW189 in healthy volunteers when given multiple doses.

DETAILED DESCRIPTION:
This is a phase 1b study. Written informed consent will be obtained from each study participant before any study-specific procedures or assessments are done.

At various time points noted below, pharmacokinetic (PK) blood sampling will be performed on study participants.

Throughout the study the investigator will be assessing adverse events and concomitant medication.

On-Study/On-Interventions Evaluations/procedures: Participants will arrive at the Phase 1 unit after fasting a minimum of 10 hours, for admission into the unit and will undergo procedures:

* Medical and medication histories
* Infection screen
* Body temperature
* Vital signs (blood pressure and heart rate)
* Physical examination and weight
* Neurological exam
* Safety laboratory tests (blood and urine)
* Urine pregnancy test (females only)
* Alcohol screening (Breathalyzer)
* Urine drug screen
* Hepatitis B, C and HIV screening
* Randomize: Only participants who meet eligibility requirements will be randomized into the study.

Day 1 - Dosing: A light breakfast will be given prior to dosing. Participants will have the following tests/procedures performed at various time points during the day following confirmation of eligibility.

* 8 electrocardiograms (ECG)
* 8 vital signs (blood pressure and heart rate)
* 1 body temperature
* 12 PK Blood draws
* 2 study drug administrations

Day 2: A light breakfast will be given prior to dosing.

* 8 ECGs
* 8 vital signs (blood pressure and heart rate)
* 1 body temperature
* 1 PK blood draw
* 2 study Drug administration

Day 3: Participants will fast for a minimum of 10 hours. Water is allowed. A Light breakfast will be given before dosing

* 1 safety laboratory tests (blood and urine)
* 1 ECG
* 2 vital signs (blood pressure and heart rate)
* 1 body temperature
* 1 PK blood draw
* 1 neurological examination
* 2 study drug administrations

Day 4: A Light breakfast will be given before dosing

* 2 vital signs (blood Pressure and heart rate)
* 1 body temperature
* 1 PK blood draw
* 2 study drug administrations

Day 5: A Light breakfast will be given before dosing

* 1 ECG
* 2 vital signs (Blood Pressure and heart rate)
* 1 body temperature
* 12 PK blood draw
* 2 study drug administration

Day 6: Participants will fast for a minimum of 10 hours. Water is allowed. A Light breakfast will be given

* 1 safety laboratory test (blood and urine)
* 1 vital sign (Blood pressure and heart rate)
* 1 body temperature
* 1 neurological examination
* 2 PK blood draw

Day 7: A light breakfast will be provided

* 1 vital sign
* 1 body temperature
* 1 PK blood draw

Day 8 (Discharge): Participants will fast for a minimum of 10 hours. Water is allowed. A light breakfast will be offered

* 1 safety laboratory test (blood and urine)
* 1 ECG
* 1 vital sign (blood pressure and heart rate)
* 1 body temperature
* 1 physical examination including weight
* 1 neurological examination

  2 Week Follow-up Visit: Participants will fast for a minimum of 10 hours. Water is allowed.

during this visit participants will have the following tests and procedures performed:

* 1 safety laboratory test (blood and urine)
* 1 ECG
* 1 vital sign (blood pressure and heart rate)
* 1 body temperature

6-8 Week Follow-up Phone Call: Participants will be asked about any adverse events and any medications they may be taking.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and capacity to give informed consent
* Is in good health
* Weights 50.0 - 120.0 kg
* Not pregnant
* Must agree to use birth control for 1 week after the last day of study drug administration
* Willingness to comply with protocol requirements, including fasting, alcohol and nicotine restrictions, during the study and is available to complete the study
* Adequate forearm vein access
* No significant dietary restrictions
* Must not have donated blood, platelets, or any other blood components 30 days, or plasma 60 days, prior to consenting. Must also agree not to donate blood, platelets, or any other blood components for 8 weeks after the last dose of study drug

Exclusion Criteria:

* Lactating or is pregnant
* severe ischemic heart disease or congestive heart failure
* Heart attack within the previous 2 years;
* history of stroke or cardiomyopathy;
* significant liver or kidney disease;
* diabetes;
* history of any autoimmune disorder; or a history of chronic infections
* a history of cancer
* has received antibiotic treatment or has undergone a surgical procedure within 30 days of Day 1
* has a history of Hepatitis C, Hepatitis B or tuberculosis (TB)
* has a history of Human Immunodeficiency Virus (HIV)
* a history of alcohol or drug use within the twelve months prior to study drug administration
* has used any immunosuppressants or chronic anti-inflammatory drugs medication including prescription medication, over-the-counter medication, health/herbal supplement or vitamin by any route of administration within 7 days of Day 1
* has donated blood within 30 days of consenting or has donated plasma within 60 days of consenting
* has participated in a clinical trial of an immunosuppressive drug within 6 months of Day 1
* has received an investigational drug, used an investigational device or received an investigational medical procedure within 60 days of Day 1, or concurrent with participation in this study
* has participated in any observational studies, experimental studies of non-investigational drugs, devices, or medical procedures within 30 days of Day 1, or concurrent with participation in this study
* has participated in a previous trial with TT301/MW189
* has a history of unexplained syncope or fainting from the collection of blood; i.e., autonomic dysfunction.
* Lack of ability to understand verbal and/ or written English
* had significant trauma or surgical procedure within 1 month prior to Screening.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda J. Van Eldik, PhD, Study Chair — University of Kentucky; Jeffrey T. Guptill, MD, MA,MHS, Principal Investigator — Duke University
Locations (1):
- Duke Clinical Research Unit 40 Duke Medicine Circle, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Van Eldik LJ, Sawaki L, Bowen K, Laskowitz DT, Noveck RJ, Hauser B, Jordan L, Spears TG, Wu H, Watt K, Raja S, Roy SM, Watterson DM, Guptill JT. First-in-Human Studies of MW01-6-189WH, a Brain-Penetrant, Antineuroinflammatory Small-Molecule Drug Candidate: Phase 1 Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Studies in Healthy Adult Volunteers. Clin Pharmacol Drug Dev. 2021 Feb;10(2):131-143. doi: 10.1002/cpdd.795. Epub 2020 Apr 7. PMID 32255549

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - TT301/MW189: TT301/MW189 0.075 mg/kg IV (or matched placebo). Each subject will receive 1 dose level of study drug twice daily (bid) on Days 1 through 5, inclusive
  Cohort 1 - TT301/MW189: 0.075 mg/kg IV twice daily on Days 1 through 5
- Cohort 2 -TT301/MW189: TT301/MW189 0.15 mg/kg IV (or matched placebo). Each subject will receive 1 dose level of study drug twice daily (bid) on Days 1 through 5, inclusive
  Cohort 2- TT301MW189: 0.15 mg/kg IV twice daily on Days 1 through 5
- Cohort 3- TT301/MW189: TT301/MW189 0.25 mg/kg IV (or matched placebo). Each subject will receive 1 dose level of study drug twice daily (bid) on Days 1 through 5, inclusive
  Cohort 3 - TT301/MW189: 0.25 mg/kg IV twice daily on Days 1 through 5
- Cohort 4- TT301/MW189: TT301/MW189 0.30 mg/kg IV (or matched placebo). Each subject will receive 1 dose level of study drug twice daily (bid) on Days 1 through 5, inclusive
  Cohort 4 - TT301/MW189: 0.30 mg/kg IV twice daily on Days 1 through 5
Period: Overall Study
Arm/Group | Placebo | Cohort 1 - TT301/MW189 | Cohort 2 -TT301/MW189 | Cohort 3- TT301/MW189 | Cohort 4- TT301/MW189
Started | 9 | 6 | 6 | 6 | 8
Completed | 6 | 6 | 6 | 6 | 4
Not Completed | 3 | 0 | 0 | 0 | 4
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: One subject who was enrolled and assigned to the placebo arm was withdrawn from the study prior to beginning the intervention. This subject is excluded from analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cohort 1 - TT301/MW189 | Cohort 2 -TT301/MW189 | Cohort 3- TT301/MW189 | Cohort 4- TT301/MW189 | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 8 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (6.7) | 32.4 (5.9) | 31.6 (6.2) | 34.5 (7.4) | 30.5 (10.9) | 33.3 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 4 | 1 | 4 | 15
  Male | 3 | 5 | 2 | 5 | 4 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 1 | 3
  Not Hispanic or Latino | 7 | 6 | 5 | 6 | 7 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 1 | 3 | 5 | 17
  White | 3 | 1 | 2 | 2 | 3 | 11
  More than one race | 1 | 1 | 3 | 0 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 6 | 6 | 8 | 34
Height [Mean (Standard Deviation); unit: cm] | 165.8 (6.7) | 171.6 (8.7) | 164.0 (11.1) | 170.9 (10.5) | 173.1 (8.4) | 169.1 (9.7)
Weight [Mean (Standard Deviation); unit: kg] | 74.5 (6.1) | 70.5 (9.1) | 75.2 (6.3) | 85.5 (20.5) | 86.4 (12.7) | 78.6 (12.8)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.1 (1.9) | 24.1 (3.8) | 28.1 (2.7) | 29.1 (5.7) | 28.8 (3.8) | 27.5 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Events
Description: The number of participants who experienced serious adverse events.
Time Frame: 4 weeks
Population: One subject randomized to the Placebo Group was withdrawn prior to receiving the study drug. Consequently, this subject is excluded from this safety analysis. As the remaining 8 subjects in the Placebo Group and all 8 subjects in Cohort 4 received an intervention they are included in safety outcomes.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort 1 - TT301/MW189 | Cohort 2 -TT301/MW189 | Cohort 3- TT301/MW189 | Cohort 4- TT301/MW189
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 8
Participants | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Treatment-Emergent Adverse Events
Description: The number of participants who experienced treatment-emergent adverse events (TEAEs). A TEAE is defined as an adverse event that started during the treatment period.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort 1 - TT301/MW189 | Cohort 2 -TT301/MW189 | Cohort 3- TT301/MW189 | Cohort 4- TT301/MW189
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 8
Participants | 5 | 6 | 4 | 6 | 6

3. Secondary Outcome: Pharmacokinetics - Cmax
Description: Maximum observed concentration in plasma.
Time Frame: 5 days
Population: Pharmacokinetic parameters for TT301/MW189 can not be analyzed in the placebo group, as they did not receive the study drug. Although 8 subjects were enrolled in Cohort 4 and are included in the safety analyses, only 4 completed sampling for PK parameters at all timepoints.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Cohort 1 - TT301/MW189 | Cohort 2 -TT301/MW189 | Cohort 3- TT301/MW189 | Cohort 4- TT301/MW189
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 4
ng/ml |  | 227 (80.5) | 347 (86.8) | 609 (180) | 750 (235)

4. Secondary Outcome: Pharmacokinetics - Tmax
Description: Time to maximum concentration
Time Frame: 5 days
Population: Tmax was not measured for any group.
Arm/Group | Placebo | Cohort 1 - TT301/MW189 | Cohort 2 -TT301/MW189 | Cohort 3- TT301/MW189 | Cohort 4- TT301/MW189
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Pharmacokinetics - AUC
Description: Area under the concentration-time curve
Time Frame: 5 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Placebo | Cohort 1 - TT301/MW189 | Cohort 2 -TT301/MW189 | Cohort 3- TT301/MW189 | Cohort 4- TT301/MW189
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 4
ng*h/ml |  | 362 (123) | 639 (220) | 1225 (474) | 1525 (458)

6. Secondary Outcome: Pharmacokinetics - T1/2
Description: Terminal half-life (T1/2)
Time Frame: 5 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | Cohort 1 - TT301/MW189 | Cohort 2 -TT301/MW189 | Cohort 3- TT301/MW189 | Cohort 4- TT301/MW189
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 4
hours |  | 8.5 (3.4) | 8.5 (3.7) | 8.8 (2.8) | 9.1 (2.8)

7. Secondary Outcome: Pharmacokinetics - Kel
Description: Elimination rate constant
Time Frame: 5 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h^-1
Arm/Group | Placebo | Cohort 1 - TT301/MW189 | Cohort 2 -TT301/MW189 | Cohort 3- TT301/MW189 | Cohort 4- TT301/MW189
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 4
h^-1 |  | 0.090 (0.029) | 0.093 (0.034) | 0.085 (0.028) | 0.081 (0.022)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Assessment was systematic. Safety and tolerability were assessed by clinical observation, lab tests and spontaneous reporting by subjects. Placebo group: 9 subjects were randomized,1 subject withdrew prior to starting the intervention. As this subject did not receive intervention, safety data are reported only for the remaining 8 subjects. Cohort 4: 8 subjects were randomized, only 4 completed all timepoints. As all 8 subjects received study drug, safety data are reported for all 8.
Arm/Group | Placebo | Cohort 1 - TT301/MW189 | Cohort 2 -TT301/MW189 | Cohort 3- TT301/MW189 | Cohort 4- TT301/MW189
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 5/8 | 6/6 | 4/6 | 6/6 | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | Cohort 1 - TT301/MW189 (N=6) | Cohort 2 -TT301/MW189 (N=6) | Cohort 3- TT301/MW189 (N=6) | Cohort 4- TT301/MW189 (N=8)
Phlebitis (Vascular disorders) | 0 | 3 | 2 | 4 | 2
Diastolic Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Pain in Extremety (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Contact Dermatitits (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 2
Infusion-Site Pain (General disorders) | 0 | 1 | 1 | 0 | 1
Infusion-Site Erythema (General disorders) | 0 | 1 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 1 | 0
Peripheral Swelling (General disorders) | 0 | 0 | 0 | 1 | 0
Infusion-Site Phlebitis (General disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 2 | 0 | 0 | 3
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 2
Parasthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Abdominal Pain, Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Sensitivity of Teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
ECG T-Wave Inversion (Investigations) | 0 | 1 | 1 | 0 | 0
Increased Blood Creatine Phosphokinase (Investigations) | 0 | 1 | 0 | 0 | 0
Decreased Hemoglobin (Investigations) | 0 | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/71/NCT02942771/Prot_SAP_000.pdf